CLINICAL TRIAL: NCT07199439
Title: Multicentre, Prospective, Post Market Observational Registry Study to Observe the Performance and Safety of the StypCel™ Device to Achieve Hemostasis During Neurosurgery
Brief Title: Post-market Clinical Follow-up Plan of StypCel™ Absorbable Hemostat
Acronym: PMCFStypcel
Status: Completed | Type: Observational
Sponsor: Medprin Regenerative Medical Technologies Co., Ltd. (Industry)
Collaborators: MDCECRO LLC (Network)
Responsible Party: Sponsor
Other Study IDs: MP-RD05-092; 270323 - 4E (Other: Latvian Ethics Committee for Clinical Research)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Neurosurgery
Keywords: bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- StypCel™ Neurosurgery Patients: This cohort includes patients undergoing neurosurgery where the StypCel™ Absorbable Hemostat is used to achieve hemostasis. The study will observe and document the effectiveness of the device in controlling bleeding during the surgery and track any subsequent complications, including infections and other adverse events, over a 6- month follow-up period

SUMMARY:
This study is a post-market clinical follow-up (PMCF) plan for the StypCel™ Absorbable Hemostat, a medical device used to control bleeding during neurosurgery. The study include 108 patients . The aim of the study is to furtherly assess the safety and performance of the device under the real-word setting

DETAILED DESCRIPTION:
The StypCel™ Absorbable Hemostat is designed to control bleeding during neurosurgical procedures. This PMCF study is an observational, multicenter study included 108 patients .Primary goal is to evaluate the device's ability to achieve hemostasis within 5 minutes during surgery. Secondary objectives include monitoring the rate of intracranial infections and other serious adverse events over 6 months. Data from the study will be collected at two-time points: 10 days and 180 days after the surgery, with follow-up assessments to monitor any delayed complications.

These summaries are written in plain language, ensuring they are accessible to non-specialists while still providing essential information about the study's objectives, methodology, and expected outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-75 years of age
* Patients requiring a hemostat device during neurosurgery.
* Patients and/or guardians agree to take part in the PMCF study and sign the Informed Consent Form.

Exclusion Criteria:

* Patients with bone defects, because it may interfere with callus formation and a possibility of cyst formation.
* StypCel™ should not be used in the control of hemorrhage from large arteries. StypCel™ should not be used as an anti-adhesion product.
* StypCel™ should not be used on the surface of non-hemorrhagic serous effusion, because in addition to the whole blood, the fluid does not react with the absorbable hemostat with satisfied hemostatic effect.
* StypCel™ is to be avoided in surgical cases requiring stuffing and packing (as is sometimes medically necessary). It may only be used in such a situation if the surgeon completely removes the device after hemostasis is achieved.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients undergoing neurosurgical procedures where the StypCel™ Absorbable Hemostat is used to control intraoperative bleeding. The population is drawn from multiple hospitals specializing in neurosurgery
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Time to Hemostasis within 5 mins | during surgery (typically within 5 minutes）
  The primary outcome is the time taken to achieve complete hemostasis at the surgical site after applying the StypCel™ Absorbable Hemostat during neurosurgery.
Time to Hemostasis | During surgery
  Time to Hemostasis within 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kaspars Auslands, Dr., Principal Investigator — Riga's East Clinical University Hospital Riga, Latvia
Locations (1):
- Riga's East Clinical University Hospital Riga, Latvia, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No